CLINICAL TRIAL: NCT03157206
Title: Peripheral Ischemia Evolution Assessed by Ultra-wide Field Angiography in Patients With Diabetic Macular Edema
Brief Title: Diabetic Retinopathy Assessed by Ultra-wide
Acronym: REGARD1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association Pour La Recherche En Vision Du Service D'Ophtalmologie De L'Hôpital (Other)
Responsible Party: Sponsor
Other Study IDs: avoph_RNI_2016-001
Record Dates: First submitted 2017-05-12; First posted 2017-05-17 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DME patients treated with aflibercept: angiography by ultrawide field

SUMMARY:
Patients with diabetic macular edema treated with aflibercept injections for visual impairment will be observed in standard care during 12 months. They will undergo visual assessments by Ultrawide Field angiography at baseline and at 12 months

DETAILED DESCRIPTION:
Diabetic retinopathy imaged by ultra wide field angiography (200°): the California (Optos, Scotland) allows ultrawide field pictures of 200° of the retina. This new imaging allows seeing beyond what was seen by the classic 7 ETDRS fields angiography:

* In pivotal studies assessing the effect of antiVEGFs on diabetic retinopathy (DR) in patients treated for diabetic macular edema (DME), ETDRS DR classification was used based on the 7 classical ETDRS field fundus photographs. However, it has been identify that antiVEGF may modified the semiology (hemorrhages, micro-aneurisms) and consecutively modify the stage of DR. There is no assessment of the regression of peripheral ischemia of the retina (non perfused retina) by angiography during an antiVEGF treatment.
* DR severity score (1) based on ETDRS classification assess the number of retinal lesions within the 7 classic retinal fields corresponding to around 30% of the total retina. It has been recently shown that peripheral lesions non visible on the classic 7 fields angiography could be predictive of progression of DR (2,3) at 4 years of follow-up independently of the initial stage of DR, HbA1C level, and could be new arguments for Laser treatment. This UWF imaging could help to understand some cases of patients with worst progression than expected, and to identify new therapeutic indications (4). These UWF pictures need to be explored in order to better characterize the severity of DR forms and probably find new therapeutics.

Impact of anti VEGF treatments on DR: pivotal studies assessing the efficacy of ranibizumab on DME explored also the effect of antiVEGFs on DR. One of the secondary endpoints of RISE and RIDE (5) studies, comparing the effect of ranibizumab 0.3mg versus 0.5mg versus sham injections, was the rate of new proliferative DR (PDR). This rate was of 33.8% in the sham group versus 11% in the treated group at 2 years of follow-up.

In Protocole I (6), the DRCRnet, found a 2 times lower risk to evolve toward PDR in case of ranibizumab treatment versus sham (7).

VIVID and VISTA showed at least 2 ETDRS steps improvement of DR for 30% of patients treated by aflibercept versus 8.2% to 15.6% at 2 years in the sham group.

It would be very interesting to have complementary data on improvement and worsening of DR under antiVEGF treatment with an angiographic analysis of the retinal periphery perfusion on larger field of the fundus than we usually have, and instead of color fundus photographs usually available in pivotal study to assess DR severity.

The purpose of this study is to characterize at one year the effect of aflibercept used for DME treatment on retinal periphery assessed by UWF angiography instead of the classic 7 ETDRS fields in order to quantify ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥ 18 years
* type 1 or type2 diabetes mellitus
* patients with at least 1 eye with best corrected visual acuity (BCVA) between 24 and 78 ETDRS letters due to center-involved diabetic macular edema (DME). DME was defined by a central retinal thickness (CRT) >300µm and the loss of foveal pit on SD-OCT
* Aflibercept treatment administred
* Afilliated to social security scheme
* agree to participate

Exclusion Criteria:

* History of treatment with any anti-VEGF agents within 12 months prior to inclusion
* Application of any intra-vitreal treatment within 12 months prior to inclusion
* Any aflibercept contraindication
* History of panretinal photocoagulation laser (PRP)
* Proliferative diabetic retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients (type 1 or 2) over 18 years of age with mild to severe non proliferative diabetic retinopathy and diabetic macular edema
Sampling Method: Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-07-18 (Estimated); Study Completion 2020-09-18 (Estimated)

PRIMARY OUTCOMES:
AntiVEGF effects on best visual acuity | 12 months
  Retinian peripheral ischemia decrease

CONTACTS AND LOCATIONS:
Locations (1):
- Giocanti-Auregan, Bobigny, France

IPD SHARING:
Plan to Share IPD: Undecided